CLINICAL TRIAL: NCT05404607
Title: Comparative Effects of Fascial Distortion Model With and Without Neuromuscular Inhibition Technique on Pain, Range of Motion and Quality of Life in Patients With Piriformis Syndrome
Brief Title: Effects of Fascial Distortion Model With and Without Neuromuscular Inhibition in Patients With Piriformis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0120
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Piriformis Syndrome
Keywords: integrated neuromuscular inhibition technique; muscle energy technique; piriformis syndrome; positional release technique; fascial distortion model
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial distortion method with neuromuscular inhibition technique (Experimental): 27 participants will receive the fascial distortion method followed by the neuromuscular inhibition technique for trigger points. After this, neural mobilization will be given as stander treatment.
  Interventions: Other: Fascial distortion method with neuromuscular inhibition technique
- Fascial distortion method (Active Comparator): Fascial distortion will be applied to 27 participants where the tip of the thumb worms its way through the peripheral tissue until it rests on the distortion. Force is focused directly on the most painful spot until the provider feels like a button-slipping-into-a-buttonhole. After this, neural mobilization will be given as a stander treatment.
  Interventions: Other: Fascial distortion method

INTERVENTIONS:
Other: Fascial distortion method with neuromuscular inhibition technique — 27 participants will receive FDM with INIT followed by neural mobilization for a total of 20 to 30 minutes, 3 times per week on alternate days for 6 weeks.
  Arms: Fascial distortion method with neuromuscular inhibition technique
Other: Fascial distortion method — 27 participants will receive FDM followed by neural mobilization for a total of 20 to 30 minutes, 3 times per week on alternate days for 6 weeks.
  Arms: Fascial distortion method

SUMMARY:
The aim of study will be to find the effects of fascial distortion model (FDM) with and without the Integrated neuromuscular inhibition technique (INIT) in piriformis syndrome.

DETAILED DESCRIPTION:
Piriformis syndrome is a misdiagnosed cause of sciatica leg or buttock pain and disability. The male and female incidence ratio of PS is 6.1. The fascial distortion model is a targeted manual technique and decodes categorized manual gestures (pain-related body language) to 6 pathophysiological mechanisms involved in the etiology of pain. Integrated neuromuscular inhibition technique(INIT) is a combination of muscle energy technique(MET) and positional release technique(PRT).

All previous studies in which integrated neuromuscular inhibition technique(INIT) and fascial distortion model(FDM) has been performed on different muscles of the body has shown greater improvement as compared to other techniques. Comparative effects of fascial distortion model with integrated neuromuscular inhibition technique and fascial distortion model on Piriformis Syndrome has not been addressed yet. There is very limited data available on this protocol. Therefore, this study aims to compare the effects of facial distortion model with and without integrated neuromuscular inhibition technique.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral buttock pain and radiculopathy due to spasms of the piriformis muscle or sciatic nerve compression.
* Aggravate buttock pain in sitting and limited SLR.
* Patient with Freiberg test positive.
* Patient with FAIR test positive.
* Patient with positive Pace test.
* Patient with positive Beatty's maneuver.

Exclusion Criteria:

* Lumbar spinal pathology and recent injury around the hip, sacroiliac joint, or lumbar spine.
* Patient with a positive Faber test
* SIJ Pathology like SIJ dysfunction, innominate anterior or posterior rotation dysfunction, etc.
* Deep gluteal syndrome.
* Recent surgery like hip arthroplasty, surgical emplacement of a gluteal implant (buttock prosthesis); lip sculpture (fat transfer and liposuction); and body contouring (surgery and lip sculpture).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Sciatica bothersomeness Index for sciatica | 6th week
  It is a composite score of four questions (each score ranging from 0-6) that include elements of leg pain and sensory and motor disturbances.
Short Form Health Survey (SF-36) questionnaire for quality of life | 6th week
  It is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions.
Goniometer for range of motion | 6th week
  It is a tool used to measure range of motions of different joints

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- GOVT Eye Cum General Hospital Gojra (THQ), Gojra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danazumi MS, Yakasai AM, Ibrahim AA, Shehu UT, Ibrahim SU. Effect of integrated neuromuscular inhibition technique compared with positional release technique in the management of piriformis syndrome. J Osteopath Med. 2021 May 31;121(8):693-703. doi: 10.1515/jom-2020-0327. PMID 34049428
- [Background] Hopayian K, Danielyan A. Four symptoms define the piriformis syndrome: an updated systematic review of its clinical features. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):155-164. doi: 10.1007/s00590-017-2031-8. Epub 2017 Aug 23. PMID 28836092
- [Background] 9. Ahmed MAA. Dexamethasone Magnesium Sulfate as an Adjuvant to Local Anesthetics in the Ultra-Sound Guided Injection of Piriformis Muscle for the Treatment of Piriformis Syndrome. The Open Anesthesia Journal. 2020;14(1).
- [Background] 10. Bose G, Dusad G. Effect of reciprocal inhibition and post isometric relaxation; types of muscle energy technique in piriformis syndrome-a comparative study. EJPMR; 2018.
- [Background] Park JC, Shim JH, Chung SH. The effects of three types of piriform muscle stretching on muscle thickness and the medial rotation angle of the coxal articulation. J Phys Ther Sci. 2017 Oct;29(10):1811-1814. doi: 10.1589/jpts.29.1811. Epub 2017 Oct 21. PMID 29184293
- [Background] Aquino-Jose VM, Blinder V, Johnson J, Havryliuk T. Ultrasound-guided trigger point injection for piriformis syndrome in the emergency department. J Am Coll Emerg Physicians Open. 2020 Jun 24;1(5):876-879. doi: 10.1002/emp2.12153. eCollection 2020 Oct. PMID 33145535
- [Background] Fishman LM, Wilkins AN, Rosner B. Electrophysiologically identified piriformis syndrome is successfully treated with incobotulinum toxin a and physical therapy. Muscle Nerve. 2017 Aug;56(2):258-263. doi: 10.1002/mus.25504. Epub 2017 Apr 2. PMID 27935076
- [Background] Han SK, Kim YS, Kim TH, Kang SH. Surgical Treatment of Piriformis Syndrome. Clin Orthop Surg. 2017 Jun;9(2):136-144. doi: 10.4055/cios.2017.9.2.136. Epub 2017 May 8. PMID 28567214
- [Background] 16. Kale A, Basol G, Kuru B, Gundogdu E, Mat E, Yildiz G, et al. Laparoscopic Surgical Approach for the Treatment of Pelvic Piriformis Syndrome. Authorea Preprints. 2020.
- [Background] Hogan E, Vora D, Sherman JH. A minimally invasive surgical approach for the treatment of piriformis syndrome: a case series. Chin Neurosurg J. 2020 Mar 30;6:8. doi: 10.1186/s41016-020-00189-y. eCollection 2020. PMID 32922937
- [Background] 18. Danazumi MS, Yakasai AM, Ibrahim SU. Effect of integrated neuromuscular inhibition technique in the management of piriformis syndrome: a case report. Middle East Journal of Rehabilitation and Health Studies. 2020;7(2).
- [Derived] Aroob Z, Bashir MS, Noor R, Ikram M, Ramzan F, Naseer A, Sabir N. Comparative effects of fascial distortion model with and without neuromuscular inhibition technique on pain, range of motion and quality of life in patients with piriformis syndrome. Disabil Rehabil. 2025 May;47(9):2378-2383. doi: 10.1080/09638288.2024.2395456. Epub 2024 Sep 3. PMID 39224057